CLINICAL TRIAL: NCT00610597
Title: Study of T Cell Phenotype Activation Pathway in Human Alcoholic Liver Disease
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Olivier Le Moine, MD, PhD, Erasme University Hospital
Other Study IDs: AL-ALD; AL-ALD
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Alcoholic Liver Disease; Chronic Hepatitis C Virus
Keywords: liver; alcohol; lymphocyte
MeSH Terms: conditions — Liver Diseases, Alcoholic; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and peripheral blood mononuclear cell culture medium.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: alcoholic liver disease
- 2: chronic hepatitis C virus infection

SUMMARY:
Alcoholic liver disease is characterized by circulating T cell activation and liver T cell infiltration but their phenotype is poorly studied. The aim of the study is to test the hypothesis that the (CD4+ T cell secreting Interleukin-17) Th17 pathway is involved in alcoholic liver disease.

DETAILED DESCRIPTION:
Consecutive patients undergoing transjugular liver biopsies for alcoholic liver disease or hepatitis C virus infection will be included in the study to measure plasma cytokines levels, peripheral blood mononuclear cells cytokine release and liver T cell infiltrates.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol excess intake and suspected liver disease
* Alcohol excess intake and clinical liver cirrhosis
* chronic hepatitis C virus infection and suspected liver disease
* chronic hepatitis C virus infection and clinical liver cirrhosis

Exclusion Criteria:

* bacterial or fungal infection
* immunosuppressive treatment
* other causes of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of Erasme University Hospital
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lemmers, MD, Principal Investigator — Erasme Hospital, Gastroenterology Dpt
Locations (1):
- Hopital Erasme - Dpt of Gastroenterology, Brussels, Belgium

REFERENCES:
- [Derived] Lemmers A, Moreno C, Gustot T, Marechal R, Degre D, Demetter P, de Nadai P, Geerts A, Quertinmont E, Vercruysse V, Le Moine O, Deviere J. The interleukin-17 pathway is involved in human alcoholic liver disease. Hepatology. 2009 Feb;49(2):646-57. doi: 10.1002/hep.22680. PMID 19177575